CLINICAL TRIAL: NCT00699036
Title: Rosiglitazone Versus Rosiglitazone and Metformin (Avandamet) Versus Combination Rosiglitazone and Losartan in the Treatment of Nonalcoholic Steatohepatitis (NASH). A Prospective, Open-Label, Randomized Trial
Brief Title: Rosiglitazone Versus Rosiglitazone and Metformin Versus Rosiglitazone and Avandia in the Treatment of Nonalcoholic Steatohepatitis (NASH)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Dawn M. Torres, MD. Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2007.066
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease
Keywords: nonalcoholic steatohepatitis (NASH); fatty liver; insulin resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Insulin Resistance | interventions — Rosiglitazone; Metformin; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): avandia
  Interventions: Drug: avandia
- 2 (Experimental): avandia plus metformin
  Interventions: Drug: avandia; Drug: metformin
- 3 (Experimental): avandia plus losartan
  Interventions: Drug: avandia; Drug: losartan

INTERVENTIONS:
Drug: avandia — 4 mg twice daily
Drug: metformin — 500 mg twice daily for 48 weeks
  Arms: 2
Drug: losartan — losartan 50 mg once daily
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy of rosiglitazone alone compared with rosiglitazone plus metformin or rosiglitazone plus losartan in the treatment of biopsy proven nonalcoholic steatohepatitis (NASH). This study was designed to answer the question: are there differences in the efficacy (as measured by histopathology and insulin resistance) of three different therapeutic modalities used to treat NASH?

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-70 years old
2. Negative urine pregnancy test in females
3. History of elevated liver associated enzymes (ALT > 40)
4. Liver biopsy within 1 year of screening in this study that shows histopathologic findings consistent with NASH

Exclusion Criteria:

1. ALT greater than three times normal
2. NYHA class 3 or 4 heart failure
3. Any congestive heart failure patient on insulin
4. Patients on one of the 3 study drugs within the past 3 months prior to enrollment
5. Alcohol consumption >20 gm/day in a female and > 30 gm/day in a male
6. Evidence of co-existent chronic liver disease to include viral hepatitis, Wilson's disease, autoimmune hepatitis, hemochromatosis, primary biliary cirrhosis, or primary sclerosing cholangitis
7. Serum creatinine on initial screening of greater than 1.4
8. Known hypersensitivity to rosiglitazone, metformin, or losartan
9. Known history of diabetic ketoacidosis
10. Female that is breastfeeding
11. Insulin dependent diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
liver biopsy histologic improvement | end of study

SECONDARY OUTCOMES:
serum transaminases | throughout study (ongoing)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Torres, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States